CLINICAL TRIAL: NCT00273221
Title: Combined Phacoemulsification and Glaucoma Implant Surgery Versus Combined Phacoemulsification and Trabeculectomy: A Randomized Controlled Trial
Brief Title: Combined Phacotube vs Phacotrabeculectomy:A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB-A/05/196
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Glaucoma; Cataract
Keywords: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Trabeculectomy; Phacoemulsification

INTERVENTIONS:
Procedure: Glaucoma Implant Surgery
Procedure: trabeculectomy
Procedure: phacoemulsification

SUMMARY:
The aim of this study is to compare the effectiveness and safety of combined phacoemulsification, posterior chamber intraocular lens implantation , trabeculectomy (phacotrabeculectomy) with phacoemulsification, intraocular lens implantation and glaucoma drainage device(phacotube) in the early and intermediate control of intraocular pressure(IOP) in patients with primary open angle and angle closure glaucoma.

DETAILED DESCRIPTION:
Studies have pointed out racial differences in the outcome of conventional filtration surgery. Glaucoma drainage implants have been found to do well in Asian eyes but no randomized controlled trial is available to support this claim. Objectives: It is the aim of this study to compare the effectiveness and safety of combined phacoemulsification, posterior chamber intraocular lens implantation , trabeculectomy (phacotrabeculectomy) versus phacoemulsification, intraocular lens implantation and glaucoma drainage device(phacotube) in the early and intermediate control of intraocular pressure(IOP) in patients with primary open angle and angle closure glaucoma. The secondary objective is to look into the post-operative complications encountered in phacotrabeculectomy and phacotube including the additional interventions (laser suture lysis, bleb needling, antimetabolite injections, etc.) applied in both procedures being studied Study Design. Randomized controlled trial. Methods. A total of 50 Asian subjects, 21 years old and above diagnosed with primary open/angle closure glaucoma, inadequately controlled by laser and medical treatment, with significant cataract and no previous eye surgery will be randomized to two types of combined procedures, phacotrabeculectomy and phacotube. Primary outcome measure is intraocular pressure and secondary outcome measures will be visual acuity, anterior chamber depth, visual field stability or progression, glaucoma medication requirement, operative and post-operative complications and additional, secondary interventions(e.g. laser suture lysis, bleb needling, 5-FU injections, anterior chamber reformation). All subjects will be followed up for a period of 1 year.This trial may define the role of GDI as a primary surgical option for Asian patients and the first randomized clinical trial in Asia to compare two combined procedures for glaucoma and cataract namely phacotrabeculectomy and phaco-glaucoma drainage implant surgery.﷡

ELIGIBILITY:
Inclusion Criteria:

Ø 21 years old and above Ø Primary Open Angle Glaucoma with Shaffer grade 2 or better for 360 degrees Ø Primary Angle Closure Glaucoma (occludable angles +/- PAS) Ø Inadequate IOP control despite maximum medical treatment (using at least 2 types or more antiglaucoma medications) and/or laser treatment in the presence of glaucomatous optic neuropathy on optic nerve head evaluation and corresponding visual field findings Ø Visually significant cataract with visual acuity of less than or equal to 6/12 Ø No corneal disease Ø Willing to be followed up for 1 year duration post-operatively Ø Informed consent

Exclusion Criteria:

* Ø Secondary Glaucoma (Uveitic, Neovascular, traumatic, Iridocorneal Endothelial Syndrome); Congenital Glaucoma Ø Severe ocular disease like Proliferative Diabetic Retinopathy, Age-related Macular Degeneration Exudative type Ø Prior intraocular surgery(in the study eye) Ø Patients with small central island and temporal field remaining on perimetry Ø One-eyed patients or fellow eye with visual acuity of counting fingers (CF) or worse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Study Completion 2006-07 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure(IOP).

SECONDARY OUTCOMES:
visual acuity,anterior chamber depth,visual field, glaucoma medication requirement, operative and post-operative complications and additional interventions(e.g.laser suture lysis, bleb

CONTACTS AND LOCATIONS:
Overall Officials: Paul TC Chew, A/Prof, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, 5 Lower Kent Ridge Road, Singapore